CLINICAL TRIAL: NCT07133334
Title: Evaluation and Comparison of the Benefits of Routine vs Shampoo Alone During 4 Weeks of Treatment and 12 Weeks Remanence n Subjects With Moderate to Severe Dandruff
Brief Title: Evaluation and Comparison of the Benefits of Routine vs Shampoo Alone During 4 Weeks Treatment and 12 Weeks Remanence
Status: Active, not recruiting | Type: Observational
Sponsor: Vichy Laboratoires (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Other Study IDs: VCY 24-011
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Dandruff
MeSH Terms: conditions — Dandruff | interventions — selenium disulfide; piroctone olamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine Dercos: Shampoo + conditionner
  Interventions: Other: Selenium disulfide; Other: Piroctone olamine
- Shampoo alone Dercos: Shampoo
  Interventions: Other: Selenium disulfide

INTERVENTIONS:
Other: Selenium disulfide — 1% SeS2
Other: Piroctone olamine — 0.5% piroctone olamine
  Groups: Routine Dercos

SUMMARY:
The goal of this study is to to evaluate and compare the efficacy of the routine "Shampoo + Conditioner " versus " Shampoo alone" immediately after application and after 1 week, 2 weeks, 3 weeks, 4 weeks (treatment phase) and 5 weeks, 8 weeks, 10 weeks and 12 weeks after applications stop (remanence phase) on subjects with moderate to severe dandruff.

Participants will:

Apply investigationnal products 3 time a week during 4 weeks and neutral or investigational products 3 time a week during 12 weeks Visit the center 9 times during the study for evaluations Keep a diary of their discomfort and the number of times they use the investigational products

DETAILED DESCRIPTION:
Secondary objectives:

* To evaluate and compare the Quality of Life (QoL) evolution of the routine " Shampoo and Conditioner " versus " Shampoo " alone, immediately after application and after 1, 2, 3, 4 weeks (treatment phase) and 5 weeks, 8 weeks, 10 weeks and 12 weeks after applications stop (remanence phase);
* To assess and compare the cosmetic properties of routine " Shampoo and Conditioner " versus " Shampoo " alone, immediately after application and after 1, 2, 3 and 4 weeks of use (treatment phase);
* To assess the tolerance of routine " Shampoo and Conditioner " versus " Shampoo " alone, during 4 weeks of use.

ELIGIBILITY:
Inclusion Criteria:

* At baseline: A moderate to severe level of squames: Total squames score (adherent + non-adherent) > 4 (ranging from 0 to 10) including an adherent squames score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent squames score at inclusion (groups must be equilibrating);
* Patient with hair length > 2 cm;
* Patient having received the information about the study modalities and having given his/her written consent and having signed the "informed consent form" specific for this study, in accordance with the corresponding procedure;
* Patient usually using a shampoo 2 to 3 times a week and accepting to follow this rate during the whole study period;
* Patient having stopped any possible soothing, anti-dandruff and anti-hair loss treatment (per os or topical) 2 weeks prior to study beginning D-14;
* Patient agreeing not to use any other hair product other than the ones provided for the study (till the end of study) in particular:
* no styling product (tonic, spray, lotion, foam) three days before the study visit;
* no treating haircare product (conditioner, hair mask, non-rinsed hair care product, oil,….);
* no anti-scales products (whatever the type: shampoo, treatment..);
* no hair colouring or hair bleaching within one week prior to any study visit.

Exclusion Criteria:

* Subject with psoriasis;
* Pregnancy, breast feeding, childbearing potential without adequate contraception, or irregular menstrual cycles;
* History of drug or alcohol abuse;
* History or suspicion of unreliability, poor cooperation or noncompliance with medical treatment;
* Topical treatment of the scalp with other antifungal medication or with corticosteroids in the last 3 weeks before start of the study;
* Systemic use of retinoids, erythromycin, tetracycline or any of its derivatives, trimethoprim/sulfamethoxazole, or metronidazole within 28 days before the start of the study.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol;
* Clinical signs and/or history of immunosuppression;
* Severe disease (e.g. cancer, cardiac infarct, unstable angina pectoris);
* Treatment with any other investigational drug in the 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe dandruff in Quatre-Borne in Mauritius
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dandruff evaluation (non adherent and adherent) | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
  Total score of dandruff = score of adherent and non adherent dandruff, which are 2 scales from 0 to 5 "0 is equivalent to no dandruff and 5 indicates a very large quantity of dandruff.

SECONDARY OUTCOMES:
Self-evaluation by subject of discomfort sensation (stinging, itching, burning sensation) on structured scale; | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
  Structured scale 0 to 9 (0 is equivalent to none, positive result and 9 indicates hugely, negative result)
Self-evaluation by subject of dandruff state and greasy aspect on structured scale | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
  Structured scale 0 to 9 (0 is equivalent to none, positive result and 9 indicates hugely, negative result)
Quality of life questionnaire - Scalpdex | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
  Publish questionnaire of quality of life, each item is evaluate with a 5-point scale from 0 (never, positive result) to 100 (always, negative result)
Standardized pictures of the scalp | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
Efficacy and cutaneaous acceptability | Day 0, Day 3, Week 1, Week 2, Week 3, Week 4, Week 9, Week 12, Week 14, Week 16
  Questionnaire with 5 proposition for each question: completely agree, somewhat agree, neitheir agree or disagree, somewhat disagree, completely disagree

CONTACTS AND LOCATIONS:
Overall Officials: Ashlam DOARIKA, Dr, Principal Investigator
Locations (1):
- Eurofins, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No